CLINICAL TRIAL: NCT00206024
Title: A 4-week Study to Investigate the Relationship Between Resolution of Acid-Associated Heartburn Symptoms and Dose of Esomeprazole Magnesium
Brief Title: Acid-Associated Heartburn Symptoms and Dose of Esomeprazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9612L00064
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Heartburn
MeSH Terms: conditions — Heartburn | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole magnesium (Nexium)

SUMMARY:
This is a multi-center, double-blind, parallel-group, randomized, proof of concept trial to investigate the relationship between dose of esomeprazole magnesium and acid-associated heartburn symptoms during 4 weeks of treatment. The safety and tolerability of esomeprazole magnesium in doses up to 40 mg BID will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-lactating females, aged 18 to 75 years, inclusive, with the ability to understand English and provide written informed consent
* A history of heartburn for at least 6 months
* A history of prior positive relief of heartburn symptoms from antacids or acid suppressive therapy
* A positive esophageal acid perfusion test
* At least 3 days of 'moderate' severity heartburn over the previous 7 days
* No use of any acid suppression therapy (PPI, H2RA, etc.) within 14 days of randomization

Exclusion Criteria:

* A history of gastric or esophageal surgery
* H. pylori positive
* A history of endoscopy -verified erosive esophagitis within the 16 weeks prior to randomization
* Currently taking higher than the standard approved proton pump inhibitor doses
* Historical evidence of a number of other GI, cardiovascular, pulmonary, liver, kidney, pancreatic, cerebral vascular diseases, organ transplant, or a condition requiring surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2004-11; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Sustained resolution of heartburn during the 4th week of treatment, defined as 7 consecutive days with a daily e-diary heartburn assessment of "None".

SECONDARY OUTCOMES:
Relief of heartburn during the 4th week of treatment
Cumulative daily sustained resolution rate through 4 weeks of treatment
Time to first day of the first 7-day period of sustained resolution of heartburn
Time to the first day of the first 7-day period of relief of heartburn
Percentage of subject-reported heartburn-free days through 4 weeks of treatment
Percentage of subject-reported heartburn-free nights through the 4 weeks of treatment
Safety and tolerability: adverse events, clinical laboratory tests, vital signs, physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Nexium Medical Science Director, MD, Study Director — AstraZeneca
Locations (27):
- United States (26):
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, DeLand, Florida
  - Research Site, Miami, Florida
  - Research Site, New Smyrna Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Hollywood, Maryland
  - Research Site, Attleboro, Massachusetts
  - Research Site, Hackensack, New Jersey
  - Research Site, Vineland, New Jersey
  - Research Site, Rochester, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Elkin, North Carolina
  - Research Site, Guthrie, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Christiansburg, Virginia
- Research Site, Ponce, Puerto Rico